CLINICAL TRIAL: NCT03365453
Title: Frailty Assessment in EldeRly Admitted to HoSpital to Receive Surgical or Percutaneous Procedure for Valvular Disorders Prospective Study
Brief Title: Frailty in Elderly Patients Receiving Surgical or Percutaneous Procedures for Valvular Disorders
Acronym: FRASER-VD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Maria Cecilia Hospital (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Associate Professor, University Hospital of Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1949
Record Dates: First submitted 2017-12-02; First posted 2017-12-07 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Age Problem; Aortic Valve Disease; Mitral Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- frailty evaluation (Experimental): all consecutive patients admitted to hospital for valvular disorders more than 69 years will be evaluated with several frailty and comorbidities scores.
  Interventions: Other: frailty evaluation

INTERVENTIONS:
Other: frailty evaluation — frailty and comorbidity scores

SUMMARY:
In Italy, life expectancy at birth has reached 80 years in men and 85 in women; in about 50 years, life expectancy at the age of 80 has increased by an extraordinary 61% and 55%, respectively, due to more effective therapies and lower mortality of many diseases. Yet, chronic diseases are nowadays more important, and often coexist as comorbidity or multimorbidity, depending on whether an index condition has been considered. These conditions increase the risk of death and reduce functional autonomy in the elderly and, therefore, should be carefully considered within comprehensive geriatric assessment. The epidemiology of valvular disease shows a clear trend in age-dependent, as the number of events and their incidence increases with age, and about half are concentrates over 75 years.

In addition, some observational studies in elderly patients have suggested an association between frailty and cardiovascular disease: fragility and cardiovascular disease share a common biological pathway, and cardiovascular diseases may accelerate the onset of frailty. The frailty syndrome was identified in 25% to 50% of patients with cardiovascular disease, according to the rating scale used and the population studied. Frail patients with cardiovascular disease, in particular those undergoing invasive procedures or suffering from coronary artery disease and aortic valve disease, have a much higher adverse events and complications, suggesting the need for a more accurate functional stratification and a more careful evaluation of the risk/benefit ratio of some invasive procedures.

Among the numerous tests proposed in the literature for the functional evaluation and objective measures of physical capability in elderly patient, the Short Physical Performance Battery (SPPB) and the evaluation of hand grip strength (grip strength) are those characterized by an improved prognostic ability and an easy administration.

The present study is performed to assess if SPPB and handgrip are helpful to better stratify the prognosis (all-causes death and hospital admission for all causes) in elderly patients admitted to hospital for cardiac causes.

DETAILED DESCRIPTION:
This is a prospective study. This a single centre study involving the Maria Cecilia Hospital (Ravenna, Italy).

The study is expected to enroll at least 450 consecutive patients with ≥70 years, which are admitted for:

GROUP A: severe aortic stenosis undergoing surgical aortic valve replacement GROUP B: severe aortic stenosis undergoing transcatheter valve implantation GROUP C: severe mitral regurgitation undergoing surgical repair GROUP D: severe mitral regurgitation undergoing MITRACLIP repair

In all patients, the following functional assessments will be performed before surgical/percutaneous intervention:

handgrip test (see definition below). Short Portable Mental Status Questionnaire (SPMSQ, see definition below). Short Physical Performance Battery (SPPB, see definition below). Multidimensional Prognostic Index (MPI, see definition below). The aim of the study is to assess the relationship between frailty score and prognosis

HANDGRIP (HGT). The handgrip test measures the force of contraction of the flexor muscles of the fingers through the use of a dynamometer. From literature it is known as such index correlates with the eventual malnutrition of the subject, with its capacity of recovery and functional recovery post-surgery, as well as to be in relation with age. In each patient, three measurements will be carried out. Will be taken into consideration for the study the highest value. The measurement will be performed as indicated by current guidelines, with the patient seated, with the dominant hand and the elbow flexed 90°. All medical personnel involved in the study performed a specific course to learn the proper management and execution of screening with handgrip tes and has personal experience in its proper execution.

SHORT PHYSICAL PERFORMANCE BATTERY (SPPB). The scale SPPB is a short battery of tests created to evaluate the functionality of the lower limbs. This battery is made up of 3 different sections designed to assess a balance with 3 tests: the maintenance of the position with the feet together for 10 seconds then the semi-tandem and finally tandem again for 10 seconds. The score of this section varies from a minimum of 0 if the patient is unable to maintain position with your feet together for at least 10 seconds to a maximum of 4 if he can accomplish all three tests. The second section of the test is intended to evaluate the progress of 4 linear meters and depending on the time of the performance section of the score ranges from 0 if unable, at one point if the performance has a longer duration of 8.7 seconds, for a up to 4 if he can accomplish the task in less than 4.80 sec. The third section investigates the ability of the battery to run for 5 consecutive times, getting up from a chair without using the arms in this regard that must be crossed in front of chest. Also in this case, the score ranges from 0 incapable or if the performance has a duration greater than 60 seconds, to a maximum of 4 if such performance is carried out in less than 11.20 seconds. The scores range from 0 (worst performance) to 12 (best performance).

A score between 5 and 9 shows seniors still independent, but with reduced physical performance, which can therefore be regarded as fragile and high risk, deserving of special attention and specific interventions, acts to reduce the risk of adverse consequences. Data in the literature confirm that the SPPB correlates with the risk of developing disability in mobility, in proportion to the decrease of the SPPB score, regardless of age, sex and presence of certain chronic diseases. The SPPB score then emerges as a powerful predictor of disability and mortality in the elderly population.

MULTIDIMENSIONAL PROGNOSTIC INDEX (MPI)

The Multidimensional Prognostic Index (MPI) is a prognostic tool based on a standard Comprehensive Geriatric Assessment (CGA) that predicts short- and long-term mortality in elderly subjects. The MPI includes 63 items distributed in 8 domains of CGA as follows:

Activities of Daily Living (ADL): 6 items Instrumental Activities of Daily Living (IADL): 8 items Short Portable Mental Status Questionnaire (SPMSQ): 10 items Mini Nutritional Assessement (MNA): 18 items Exton-Smith Scale (ESS): 5 items Cumulative Index Rating Scale - Comorbidity Index (CIRS-CI): 14 items Number of drugs used: 1 item Co-habitation status: 1 item On the basis of MPI values, it is possible to calculate the short- and long-term mortality risk of the older subjects and to define the severity grade of mortality risk: low, moderate and severe. Several studies showed that the prognostic accuracy of the aggregated MPI was significantly greater than the prognostic accuracy of its individual components considered singularly. Thus the multidimensional approach can be successfully used in elderly patients for both clinical and administrative purposes.

ELIGIBILITY:
Inclusion Criteria:

* age ≥70
* hospital admission for valvular disorders (severe aortic stenosis or severe mitral regurgitation) requiring surgical or percutaneous intervention

Exclusion Criteria:

* SPMSQ value ≤4
* inability to stay upright
* life expectancy <3 months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 450 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
composite endpoint of all-cause mortality and all-cause hospital admission | 1-year
  1-year cumulative incidence of all-cause mortality and all-cause hospital admission

SECONDARY OUTCOMES:
all-cause mortality | 1-year
  1-year cumulative incidence of death for all-causes
cardiac death | 1-year
  1-year cumulative incidence of cardiac death
cardiac adverse events | 1-year
  1-year cumulative incidence of cardiac death, myocardial infarction, heart failure

OTHER OUTCOMES:
cerebrovascular accident | 1-year
  1-year cumulative incidence of stroke and/or transient ischemic attack

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Campo, Principal Investigator — Azienda Ospedaliera Universitaria di Ferrara; Alberto Cremonesi, Principal Investigator — Maria Cecilia Hospital
Locations (1):
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: Undecided